CLINICAL TRIAL: NCT06243432
Title: Estrogen Receptors and HER2 Levels' Expression in Luminal Metastatic Breast Cancer: Correlation to Therapeutic Efficacy of Cycline-Dependent Kinase Inhibitors(CDK4/6) as First Line Treatment. CYCLHER Study
Brief Title: Estrogen Receptors and HER2 Levels' Expression in Luminal Metastatic Breast Cancer
Acronym: CYCLHER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5519
Record Dates: First submitted 2024-01-24; First posted 2024-02-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-10

CONDITIONS: Advanced Breast Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CYCLHER is a retrospective observational multicentric italian study aimed to evaluate the correlation between hormone receptors (HR) and HER2 immunohistochemistry (IHC) levels and treatment'response in patients affected by advanced breast cancer treated with first line CDK4/6 inhibitor plus endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yo
* Histological diagnosis of HR+/HER2- advanced breast cancer
* Immunohistochemical HER2 negative evaluation (0, 1+ or 2+ FISH-)
* Immunohistochemical expression levels of estrogen and progesterone receptors
* First line CDK4/6 inhibitor plus endocrine therapy stared up to 12/31/2020
* Signing of informed consent approved by local Ethic Committee

Exclusion Criteria:

* Absence of clinical and pathological data that would compromise the definition of the study endpoints
* HER2 positive (ICH 2+ and FISH positive or HER2 3 +) or triple negative disease
* Previous chemotherapy for treatment of metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- advanced breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Through study completion, an average of 1 year".
  PFS of HR+/HER2- breast cancer patients who received endocrine treatment plus CDK4/6 inhibitor as first line treatment for metastatic disease, categorized according to estrogen and progesterone receptor levels and HER2 expression status (HER2 0,1+ or 2+ FISH negative).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 1 year".
  ORR according to estrogen and progesterone receptor levels and HER2 expression status (HER2 0,1+ or 2+ FISH negative).
Overall survival (OS) | Through study completion, an average of 1 year".
  OS according to estrogen and progesterone receptor levels and HER2 expression status (HER2 0,1+ or 2+ FISH negative).
Incidence of Adverse Events (AEs) | Through study completion, an average of 1 year".
  AEs related to the treatment and evaluated according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico A. Gemelli - IRCCS, Rome, Italy